CLINICAL TRIAL: NCT05415150
Title: MEASUREMENT OF MARKERS OF PLATELET AGGREGATION AND INFLAMMATION IN ISCHEMIC STROKE SUBJECTS AFTER FIBRINOLYTIC/ANTI-THROMBOTIC USE. A PILOT STUDY.
Brief Title: Platelet Function in Patients With Ischemic Stroke Treated With Anti-thrombotic or Thrombolytic
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Pitchaiah Mandava, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31232
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Fibrinolytic Agents; Eptifibatide; Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Measurement of Platelet function (Experimental): Patients with ischemic stroke may be given alteplase or other thrombolytic. Additionally, patients may be given IV platelet inhibitors and subjected to thrombectomy. Platelet functions are measured after intervention.
  Interventions: Drug: Thrombolytic Agent

INTERVENTIONS:
Drug: Thrombolytic Agent — Subjects may receive one or more of the treatment options
  Other Names: eptifibatide; thrombectomy

SUMMARY:
Acute stroke afflicts nearly 700,000 patients in the US and is the number 3 cause of death. Only 2-9% of this large number is treated with t-PA if they arrive within 4.5 hours. An equally small percentage of patients with large vessel occlusion undergo thrombectomy.

The thrombectomy patients may or may not receive t-PA. Some of these patients rarely receive intravenous GPIIB/IIIa inhibitors. Many lines of evidence suggest that GP IIb/IIIa inhibitors, a class of FDA approved potent platelet inhibitors that have been used extensively along with heparin for acute coronary syndromes (heart attacks) and unstable angina (chest pain), may be safe enough to give in these circumstances.

DETAILED DESCRIPTION:
In the past we used 30% lower dose of abciximab compared to the cardiac trials and the discontinued ABESTT stroke trial. There were no symptomatic intracranial hemorrhages or thromboyctopenia in our study. Based on the safety and efficacy results (Mandava et al, Translational Stroke Research 2010), we continued its use until manufacture of this agent was stopped.

There is another compound eptifibatide (Integrilin), that is also a GP IIb/IIIa which is in use in acute coronary syndromes. Eptifibatide has been used by cardiologists since 1998. Reduced doses have been studied along with intravenous rt-PA in stroke patients [Pancioli et al 2008 and 2013].

We are proposing even smaller dose compared to Pancioli et al 2008 and 2013. The reduced dose proposed here is less than 1/10th (<10%) cardiac dose. For an 80 kg patient the cardiac dose is 244 mg (14 mg bolus followed by an infusion of 230 mg over 24 hours). The reduced dose proposed here for stroke for an 80 kilogram patient is 10 mg bolus followed by an infusion of 10 mg over 24 hours. For patients weighing more than 80 kg the maximum bolus and infusion doses will remain 10 mg each. The cardiac dose does not specify a maximum weight.

If patients are eligible to receive alteplase as standard of care, patients will be offered alteplase.

Platelet aggregation has many poorly understood complex roles in ischemic stroke. We are planning on drawing three tubes of blood in addition before and after treatment. The tubes of blood will be collected at the bedside after consent and will be coordinated with the regularly scheduled blood draw that a patient undergoes at presentation to the emergency room. The three tubes of blood will be obtained and tests available in the laboratory will be performed. The three tests are Platelet Function Assay (PFA), Verify-Now (Aspirin) and Verify-Now(Plavix).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 18 years or older
2. Anterior Circulation stroke within the last six hours
3. Posterior Circulation stroke within the last 12 hours

Exclusion Criteria:

1. Initial CT of the head suggests stroke like symptoms are not due to an ischemic stroke but a result of hemorrhage or tumor
2. Platelet count below 100,000
3. PTT greater than 75 while on treatment with heparin
4. INR greater than 2.5 while on treatment with warfarin
5. ACT>250
6. Have clinical signs and symptoms of liver failure or elevations in AST, and ALT > 3 times the normal values.
7. Creatinine greater than 2
8. Treatment team considers the patient to be at increased risk of intra-cerebral hemorrhages or systemic bleeding
9. Pre-morbid modified Rankin score >2 suggesting a functionally dependent patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Ninety day functional outcomes | Ninety days
  Modified Rankin Score

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States